CLINICAL TRIAL: NCT04638868
Title: A Head-to-head Comparison of a Novel Silicon Microsieve Device Against a Cell Surface Marker-based Platform for the Isolation of Portal Vein Circulating Tumor Cells in Pancreatic Cancer
Brief Title: Silicon Microsieve Device vs Cell Surface Marker-based Platform for the Isolation of Pancreatic Cancer CTCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/2502; 03/FY2018/P1/13-A28FY2019PFF02 (Other Grant/Funding Number: Singapore General Hospital)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Pancreatic Cancer
Keywords: Circulating Tumor Cells; Endoscopic Ultrasound; Portal vein blood sampling; Fine needle aspiration; Microsieve
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isolation of circulating tumor cells (Experimental): Both portal venous and peripheral blood will be obtained from the patient and subjected to analysis for pancreatic cancer circulating tumor cells
  Interventions: Device: Microsieve device; Device: Cell surface marker-based platform

INTERVENTIONS:
Device: Microsieve device — Both portal venous and peripheral blood will be processed through a label-free size-based silicon microsieve microfiltration device, which will isolate both epithelial-type and mesenchymal-type pancreatic cancer circulating tumor cells. Downstream mutational analyses will be performed to confirm identity of the cells.
Device: Cell surface marker-based platform — Both portal venous and peripheral blood will be processed through a cell surface marker-based platform, which contains antibodies for epithelial cell markers on pancreatic cancer circulating tumor cells. Downstream mutational analyses will be performed to confirm identity of the cells.

SUMMARY:
The study aims to compare the use of a microsieve device vs a cell surface marker-based platform for the isolation of pancreatic cancer circulating tumor cells

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs) aid prognostication of cancer by predicting the presence of microscopic metastases. This is important in pancreatic cancer, which is associated with a poor prognosis even in resectable disease, due to microscopic metastases that are not detectable on pre-operative cross-sectional imaging. In pancreatic cancer, blood is sampled from the portal circulation to overcome the "hepatic sieve" effect, where CTCs are filtered out in the capillary beds of the liver before entering the peripheral circulation. Minimally invasive blood sampling from the portal vein can now be done via endoscopic ultrasound (EUS) guidance, allowing CTC analyses to be done pre-operatively.

CTCs have traditionally been isolated in various cancers using a cell surface marker-based platform (CellSearch™). This involves the use of antibodies to identify, isolate and quantify CTCs based on presence of specific epithelial cell markers. However, CTCs are now known to undergo epithelial-mesenchymal transformation. The current epithelial cell surface marker-based method of CTC isolation is limited by its inability to detect mesenchymal-type CTCs, potentially under estimating the CTC count, affecting quantification and subsequent CTC molecular analyses.

The use of a novel silicon microsieve device will overcome these limitations. It will simplify the isolation of CTCs by its characteristic size, enable both epithelial and mesenchymal types of CTCs to be isolated and results in greater cell viability, aiding in subsequent cell culture and organoid growth.

The investigators will compare a novel silicon microsieve size-based cell filtration device against the cell surface marker label-based CellSearch™ platform for the identification of pancreatic cancer CTCs in portal venous blood obtained via an Endoscopic Ultrasound (EUS)-guided puncture. The investigators will compare the yield of epithelial-type CTCs isolated using both methods. The investigators will investigate whether the isolation of mesenchymal-type CTCs via a sized-based cell filtration device leads to a significant increase in total CTC yield.

The investigators expect our study to show that the new technique of size-based CTC isolation improves CTC yield in pancreatic cancer. This preliminary data would be crucial for future research into patient selection for neoadjuvant chemotherapy and individualized treatment from patient-specific tumor tissue, which the investigators intend to embark upon.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and older
2. All inpatients with solid pancreatic lesions referred for Endoscopic Ultrasound - Fine Needle Aspiration (EUS-FNA)
3. Solid lesions confirmed by at least a single investigational modality, mainly CT, MRI or endoscopy
4. Able to comply with the study procedure and provide informed consent.

Exclusion Criteria:

1. Presence of active bleeding
2. Presence of coagulopathy as evidenced by INR >1.5 and platelets <50,000
3. Poor patient tolerance to procedure
4. Concurrent intake of anticoagulants and thienopyridine (e.g.Clopidogrel) in patients who require antiplatelet therapy
5. Pregnancy
6. Presence of portal vein thrombus
7. Patients with liver cirrhosis and /or other structural abnormalities in the liver or the stomach

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-11-17 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of circulating tumor cells | Immediately following procedure
  The number of circulating tumor cells isolated via both methods (microsieve device and cell surface marker-based platform)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Meng Yew Tan, MBBS, Principal Investigator — Singapore General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman CG, Waxman I. EUS-guided portal vein sampling. Endosc Ultrasound. 2018 Jul-Aug;7(4):240-245. doi: 10.4103/eus.eus_28_18. PMID 30117486
- [Result] Tien YW, Kuo HC, Ho BI, Chang MC, Chang YT, Cheng MF, Chen HL, Liang TY, Wang CF, Huang CY, Shew JY, Chang YC, Lee EY, Lee WH. A High Circulating Tumor Cell Count in Portal Vein Predicts Liver Metastasis From Periampullary or Pancreatic Cancer: A High Portal Venous CTC Count Predicts Liver Metastases. Medicine (Baltimore). 2016 Apr;95(16):e3407. doi: 10.1097/MD.0000000000003407. PMID 27100430
- [Result] Catenacci DV, Chapman CG, Xu P, Koons A, Konda VJ, Siddiqui UD, Waxman I. Acquisition of Portal Venous Circulating Tumor Cells From Patients With Pancreaticobiliary Cancers by Endoscopic Ultrasound. Gastroenterology. 2015 Dec;149(7):1794-1803.e4. doi: 10.1053/j.gastro.2015.08.050. Epub 2015 Sep 2. PMID 26341722
- [Result] Christiansen JJ, Rajasekaran AK. Reassessing epithelial to mesenchymal transition as a prerequisite for carcinoma invasion and metastasis. Cancer Res. 2006 Sep 1;66(17):8319-26. doi: 10.1158/0008-5472.CAN-06-0410. PMID 16951136
- [Result] Cima I, Wen Yee C, Iliescu FS, Phyo WM, Lim KH, Iliescu C, Tan MH. Label-free isolation of circulating tumor cells in microfluidic devices: Current research and perspectives. Biomicrofluidics. 2013 Jan 24;7(1):11810. doi: 10.1063/1.4780062. eCollection 2013. PMID 24403992